CLINICAL TRIAL: NCT03799718
Title: A Phase 2 Open-label Multicenter Study to Evaluate the Safety and Efficacy of Repeated Administration of NurOwn® [Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors (NTF), MSC-NTF] Cells in Participants With Progressive MS
Brief Title: Safety and Efficacy of Repeated Administration of NurOwn (MSC-NTF Cells) in Participants With Progressive MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brainstorm-Cell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT-101-US
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis, Chronic Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NurOwn (MSC-NTF cells) (Experimental): Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors
  Interventions: Biological: NurOwn (MSC-NTF cells)

INTERVENTIONS:
Biological: NurOwn (MSC-NTF cells) — Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors

SUMMARY:
A multidose open-label study with autologous Mesenchymal Stromal Stem Cells Secreting Neurotrophic Factors (MSC-NTF cells) involving 20 participants with progressive MS at multiple investigational study sites.

DETAILED DESCRIPTION:
An open-label study with a single treatment arm involving 20 participants with progressive MS at multiple investigational study sites. After providing informed consent, participants meeting the inclusion and exclusion criteria will be randomized and approximately 4 weeks later will undergo a bone-marrow aspiration (BMA). Each participants will receive three Intrathecal cell transplantations within 16 weeks and will be followed for 12 weeks for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18 to 65 years old, inclusive, at the Screening Visit.
2. Clinical diagnosis of Progressive MS (Primary and Secondary) based on the 2017 revised MacDonald Criteria and confirmation by the Investigator that the disease has entered the progressive stage for at least 6 months prior to enrollment.
3. No evidence of clinical MS relapse or high dose pulse corticosteroid treatment within 6 months prior to screening
4. Disability status at screening with an Expanded Disability Status Scale (EDSS) 3.0-6.5, inclusive.
5. Able to walk 25 feet in 60 seconds or less.
6. Stable dose of non-excluded MS Disease Modifying Therapy for at least 6 months prior to Screening Visit (Visit 1).
7. Women of childbearing potential shall either be surgically sterile, or must agree not to become pregnant for the duration of the study. Women must be willing to undergo a serum pregnancy test at screening, and at the conclusion of the study. Participants of childbearing potential must agree to use a medically approved form of birth control (abstinence, intrauterine device (IUD), oral contraception, barrier and spermicide or hormonal implant) throughout the duration of the study and for at least 3 months following the last transplantation. For those women who are sexually active and using oral contraceptives, a second form of barrier contraception is required. Men must be willing to consistently use two forms of contraceptive if their partners are of childbearing age.
8. Capable of providing informed consent and willing and able to follow study procedures, including willingness to undergo multiple/repeated lumbar puncture.

Exclusion Criteria:

1. Prior stem cell therapy of any kind.
2. Active participation in any other MS interventional study or use of unapproved MS investigational therapy within 90 days prior to the Screening Visit (Visit 1).
3. Inability to lie flat for the duration of intrathecal cell transplantation and/or bone marrow biopsy, or inability to tolerate study procedures for any other reason.
4. History of clinically significant autoimmune disease (excluding thyroid disease) that may confound study results, in the opinion of the Investigator and the medical monitor, myelodysplastic or myeloproliferative disorder, leukemia or lymphoma, whole body irradiation, hip fracture, or severe scoliosis.
5. Any unstable clinically significant medical condition other than multiple sclerosis (e.g., within six months of Screening Visit (Visit 1), had myocardial infarction, angina pectoris, and/or congestive heart failure), treatment with anticoagulants that, in the opinion of the investigator, would compromise the safety of participants.
6. Any history of malignancy within the previous 5 years, except for non-melanoma localized skin cancers (with no evidence of metastasis, significant invasion, or reoccurrence within three years of Screening Visit (Visit 1)).
7. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value >3.0 times the upper normal limit.
8. Serum creatinine value >2.0 times the upper normal limit.
9. Positive test for Hepatitis B (HBV; surface antigen (HBsAg) and antibodies to core antigen (IgG and IgM anti-HBc)), Hepatitis C (HCV), or human immunodeficiency virus (HIV) 1 and 2.
10. Current use of immunosuppressant medication or use of such medication within 6 months of study enrollment (aside from Rituximab or other approved B-cell immunotherapy). Alemtuzumab (Lemtrada), Cladribine (NDA submitted), Natalizumab (Tysabri), S1P modulators (Gilenya) are excluded for safety reasons due to the known risk of systemic autoimmune disease, malignancy, opportunistic infections, and cardiovascular toxicity associated with these therapies, as well as theoretical effects on MSC-NTF cell homing and migration, that may be associated with Natalizumab and/or S1P modulators (Gilenya).
11. Any history of acquired or inherited immune deficiency syndrome.
12. Any history of either substance abuse within the past year, or unstable psychiatric disease according to the Investigator's judgment.
13. Pregnant women or women currently breastfeeding.
14. Subjects for whom MRI is contraindicated (i.e., have a pacemaker or other metallic implanted device, or are unable to remain in the machine for period of time needed to acquire a scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cohen, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Stanford University School of Medicine, Redwood City, California
  - The Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not meeting inclusion exclusion criteria
Units Other Than Participants: Treatments
Groups:
- NurOwn (MSC-NTF Cells): Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors NurOwn (MSC-NTF cells). Study drug was supplied in one 5 mL syringe containing 4 mL of NurOwn (MSC-NTF cells) suspension at a dose of 100-125 x106 cells for IT administration. 3 doses of NurOwn (MSC-NTF cells) were transplanted intrathecally at 8-week intervals (Day 0-1, week 8, and week 16)
Period: Overall Study
Arm/Group | NurOwn (MSC-NTF Cells)
Started | 20; 54 Treatments (20 participants underwent bone marrow aspiration. In two participants, autologous bone marrow culture failed to meet specific MSC-NTF cell product release criteria and they did not receive treatment)
Completed | 18; 53 Treatments (Of the 20 participants enrolled, 18 were treated, 17 received all three treatments and one received two treatments.)
Not Completed | 2; 1 Treatments
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are for participants with a clinical diagnosis of primary or secondary progressive MS (PPMS or SPMS) based on the 2017 revised McDonald Criteria and confirmation by the Investigator that the disease has entered the progressive stage at least 6 months prior to enrollment
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Timed 25-foot walk speed [Mean (Standard Deviation); unit: Feet/seconds] — The T25FW is a quantitative mobility and leg function performance test based on a timed 25-feet walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Baseline T25FW is the average of the two successive trials. Higher values represent better outcomes
  Feet/seconds | 2.4 (1.6)
Nine-Hole Peg Test (9HPT) [Mean (Standard Deviation); unit: Seconds] — The Nine-Hole Peg Test (9HPT) is used to measure upper extremity function in patients with various neurological diagnoses The participant is seated at a table with a container holding nine pegs and a block with 9 empty holes. On a start command, the participant picks up the nine pegs, puts them in the nine holes, and, once completed, removes them again as quickly as possible, replacing them into the container. The total time to complete the task is recorded.
  Baseline 9HPT is the average of 2 trials of dominant hand and nondominant hand. Higher values represent a worse outcome.
  Seconds | 35.2 (15.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Combined safety of all 3 intrathecal doses of NurOwn® (MSC-NTF cells) Number of participants who experienced Treatment-emergent Adverse Events during the study.
  Treatment-emergent Adverse Event is an adverse event that occurs for the first time after initiation of first treatment or if it had occurred prior to initiation first treatment, it worsens in severity after initiation of first treatment.
Time Frame: Up to 28 weeks post-first treatment
Population: The primary, secondary, and exploratory efficacy endpoints were analyzed using the modified intent to treat (mITT) and Efficacy Evaluable (EE) populations The mITT population was defined in this study as all participants who received at least 1 treatment and had at least 1 T25FW or 9-HPT assessment post baseline. Baseline was defined as the most recent assessment prior to receiving the first transplantation on Day 0, at Visit 3
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants | 18

2. Secondary Outcome: Number of Participants With 25% or Greater Improvement From Baseline in Time 25 Foot Walk (T25FW) Speed or Nine-Hole Peg Test (9-HPT)
Description: 25% or greater improvement at 28 weeks from Baseline in Time 25 Foot Walk (T25FW) speed or 9 Hole Peg Test (9-HPT).
  The T25FW is a quantitative mobility and leg function performance test based on a timed 25-feet walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. T25FW is the average of the two successive trials. Higher values represent better outcomes.
  The 9HPT is used to measure upper extremity function in patients with various neurological diagnoses. The participant is asked to pick up the nine pegs, puts them in the nine holes, and, once completed, removes them again as quickly as possible, replacing them into the container. The total time to complete the task is recorded.
  Higher values represent worse outcomes.
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: The modified intent to treat (mITT) population was defined in this study as all participants who received at least 1 treatment and had at least 1 T25FW or 9-HPT assessment post baseline. Baseline was defined as the most recent assessment prior to receiving the first transplantation on Day 0, at Visit 3
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants
  Number of Participants with 25% or greater improvement from Baseline inT25FW speed or 9-HPT | 3
  Number of Participants with <25% improvement from Baseline inT25FW speed or 9-HPT | 13
  Number of Participants with missing data at week 28 | 2

3. Secondary Outcome: Number of Participants With 25% or Greater Improvement From Baseline to Week 28 in Timed 25 Foot Walk (T25FW) Speed
Description: ≥25% improvement in T25FW speed over 28 weeks The T25FW is a quantitative mobility and leg function performance test based on a timed 25-feet walk.
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely.
  The task is immediately administered again by having the patient walk back the same distance Baseline T25FW is the average of the two successive trials. Higher values represent better outcomes
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants
  Number of participants with 25% or more improvement | 2
  Number of participants without 25% or more improvement | 12
  Number of participants with missing values at week 28 | 4

4. Secondary Outcome: Number of Participants With 25% or Greater Improvement From Baseline to Week 28 in 9-HPT
Description: The Nine-Hole Peg Test (9HPT) is used to measure upper extremity function in patients with various neurological diagnoses.
  The participant is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. On a start command when a stopwatch is started, the participant picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand.
  Baseline 9HPT is the average of 2 trials of dominant hand and nondominant hand. The higher values represent a worse outcome.
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: The mITT population was defined in this study as all participants who received at least 1 treatment and had at least 1 T25FW or 9-HPT assessment post baseline. Baseline was defined as the most recent assessment prior to receiving the first transplantation on Day 0, at Visit 3.
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants
  Number of Participants with 25% or greater improvement from Baseline to Week 28 in 9-HPT | 2
  Number of Participants with less than 25% improvement from Baseline to Week 28 in 9-HPT | 13
  Number of participants with missing values at week 28 | 3

5. Secondary Outcome: Number of Participants Who Had >5.5 in Expanded Disability Status Scale (EDSS) at Baseline, With ≥0.5 Points Improvement From Baseline to Week 28
Description: Expanded Disability Status Scale (EDSS) provides a total score on a scale that ranges from 0 (no disability) through 1 to 10 (death due to MS), in 0.5-point steps. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the sequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The higher score represents the worse outcome.
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: The mITT population was defined in this study as all participants who received at least 1 treatment and had at least 1 T25FW or 9-HPT assessment post baseline.
  Baseline was defined as the most recent assessment prior to receiving the first transplantation on Day 0, at Visit 3.
  The participants in mITT population whose EDSS Score was >5.5 at Baseline was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 10
Participants
  No of Participants with >5.5 in EDSS at Baseline with ≥0.5 Points Improvement from Baseline to Wk 28 | 3
  No of Participants with >5.5 in EDSS at Baseline with <0.5 Points Improvement from Baseline to Wk 28 | 7

6. Secondary Outcome: Number of Participants With ≥10 Points Improvement From Baseline to Week 28 in Multiple Sclerosis Walking Scale (MSWS-12)
Description: The Multiple Sclerosis Walking Scale (MSWS)-12 is a patient-reported outcome measure of the walking limitations due to MS during the past 2 weeks.
  It contains 12 questions that assess the impact of MS on different aspects of walking function and quality.
  Total administration time should be approximately 5 minutes. Activities are rated by participant from min. 1 (not at all) to max. 5 (extremely) and summed to calculate a total score using a scale from 0 to 60 (ranging from low to high impact on walking). This score is then divided by 60 and multiplied by 100 to get a score between 0 and 100 A higher score represents a worse outcome.
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants
  Number of Participants with ≥10 Points Improvement from Baseline to Week 28 in MSWS-12 | 6
  Number of Participants with <10 Points Improvement from Baseline to Week 28 in MSWS-12 | 10
  Number of Participants with missing data at week 28 | 2

7. Secondary Outcome: Number of Participants With ≥8 Letter Improvement From Baseline to Week 28 in LCLA Binocular 2.5% Contrast Level
Description: The Low contrast letter acuity (LCLA) is a leading outcome measure to assess visual disability in multiple sclerosis (MS) research Total administration time, for a typical MS patient, is approximately 10-15 minutes to complete, when testing each eye individually and binocular vision for two different contrast levels.
  The score for each chart is quantified as the number of letters identified correctly with a minimum scrore of 0 letter and a maximum score of 70 letters. The higher score represents the better outcome.
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants
  No. of participants with ≥8 Letter improvement at Week 28 in LCLA Binocular 2.5% Contrast Level | 4
  No. of Participants with <8 Letter Improvement at week 28 in LCLA Binocular 2.5% Contrast Level | 11
  Number of Participants with missing data at week 28 | 3

8. Secondary Outcome: Number of Participants With ≥ 3 Points Improvement From Baseline to Week 28 in Symbol Digit Modalities Test (SDMT) Score
Description: Symbol Digit Modalities test (SDMT) is a commonly used test to assess psychomotor speed, which measures processing speed as well as motor speed.
  It is a paper-pencil measure which requires an individual to substitute digits for abstract symbols using a reference key Scoring involves summing the number of correct substitutions within the 90 second interval (max = 110) Minimum score is 0 and maximum score 110. The higher score represents the better outcome.
Time Frame: From Baseline (pre-first treatment) to 28 weeks post-first treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 18
Participants
  Number of Participants with ≥ 3 points Improvement from Baseline to Week 28 in SDMT Score | 10
  Number of Participants with < 3 points Improvement from Baseline to Week 28 in SDMT Score | 5
  Number of Participants with missing data at week 28 | 3

9. Secondary Outcome: Change in Concentration of Vascular Endothelial Growth Factor (VEGF) Neuroprotective Biomarker From Baseline in the Cerebrospinal Fluid (CSF) 16 Weeks Following First NurOwn® Treatment
Description: Change from baseline (pre-first treatment) in the concentration of Vascular endothelial growth factor (VEGF) neuroprotective biomarker in the Cerebrospinal fluid (CSF) at 16 weeks following first NurOwn® treatment The concentration of the biomarker is measured as Picogram per milliliter (pg/ml). A higher concentration of neuroprotective biomarkers suggests a better outcome
Time Frame: From Baseline (pre-first treatment) to 16 weeks post first treatment
Population: mITT Population with data available at week 16
Measure: Geometric Mean (Inter-Quartile Range); unit: Picograms per milliliter
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 17
Picograms per milliliter | 90.17 [-9.16 to 124.80]

10. Secondary Outcome: Change in Concentration of Hepatocyte Growth Factor (HGF) Neuroprotective Biomarker From Baseline in the Cerebrospinal Fluid (CSF) 16 Weeks Following NurOwn® Treatment
Description: Change from baseline in the concentration of Hepatocyte growth factor (HGF) neuroprotective biomarker in the Cerebrospinal Fluid (CSF) at 16 weeks following the first NurOwn® treatment The concentration of the biomarker is measured as Picogram per milliliter (pg/ml). A higher concentration of neuroprotective biomarkers suggests a better outcome
Time Frame: From Baseline (pre-first treatment) to 16 weeks post first treatment
Population: mITT population with data available at week 16
Measure: Geometric Mean (Inter-Quartile Range); unit: picograms per milliliter
Arm/Group | NurOwn (MSC-NTF Cells)
Number analyzed (Participants) | 17
picograms per milliliter | 15.16 [0.2 to 19.44]

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: Adverse Events (AE) were collected over a period of 38 weeks from the time of informed consent at the screening visit through the last study visit (Visit 7 or an Early Termination visit) Treatment Emergent Adverse Events (TEAE) were collected over a period of 28 weeks from the time of the first treatment through the last study visit (Visit 7 or an Early Termination visit)
Arm/Group | NurOwn (MSC-NTF Cells)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NurOwn (MSC-NTF Cells) (N=18)
Arachnoiditis (Nervous system disorders) | 2 (2) — [1] Two participants experienced an SAE of arachnoiditis in one of three treatments (one participant with Grade 1 and one participant with Grade 3) that were considered probably related to the IT injection procedure and/or study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NurOwn (MSC-NTF Cells) (N=18)
Headache (Nervous system disorders) | 16 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (29)
Urinary tract infection (Infections and infestations) | 6 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Injection site pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Fatigue (General disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03799718/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03799718/SAP_001.pdf